CLINICAL TRIAL: NCT02957162
Title: The Effect on Endothelial Progenitor Cells (EPCs) by Statin Loading in "All Comers" With an Acute Coronary Syndrome (ACS)
Brief Title: The Effect on EPCs by Statin Loading in "All Comers" With an ACS
Acronym: ALL COMERS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 995
Record Dates: First submitted 2016-10-19; First posted 2016-11-07 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Atorvastatin; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood samples and Atorvastatin 80mg (Other): All participants are given Atorvastatin 80mg as part of their standard care. The main study intervention is blood samples at days 1-2, 3-4 and 7-8.
  Interventions: Drug: Atorvastatin; Other: Blood samples

INTERVENTIONS:
Drug: Atorvastatin
Other: Blood samples — 3-5 mls of blood is taken at baseline and 3 subsequent timepoints and processed for Endothelial Progenitor Count (EPC).

SUMMARY:
Cardiovascular disease is a major cause of morbidity and mortality worldwide. There are a number of risk factors for coronary artery disease and all to often patients admitted with an acute coronary syndrome have these comorbidities.

The main stay of treatment of such patients is to perform coronary angiography and if required coronary angioplasty.

Previous studies have shown a link between endothelial progenitor cell (EPC) count, coronary artery disease and statin therapy or loading, however these studies have excluded patients with significant comorbidities and therefore have not truly represented "real life" patients. This pilot study will assess EPC response in patients that are able to undergo coronary intervention as part of their normal clinical management under current guidelines regardless of pre-existing comorbidities. The research team believe this will allow representation of "real world" patients.

DETAILED DESCRIPTION:
This pilot study will include up to 40 patient-participants admitted into the coronary care unit of the Royal Stoke University Hospital a large and busy tertiary cardiac centre. Patient-participants will be assessed, and if deemed appropriate to undergo coronary angiography and or angioplasty will be eligible for enrolment in the study.

Following standard care angiogram / angioplasty, patient-participants will be given a minimum of 3 hours to consent to ensure that there is no delay in clinical treatment. A short information sheet will be given to the patient initially. If the patient is interested in the study, the full participant information sheet will be given. If potential patient-participants consent to study participation 3-5ml of blood will be venesected and sent for EPC analysis. That late evening atorvastatin 80mg will be given as per current national recommendations. Patient-participants will then have venesection for EPC analysis on days 1-2, 3-4 and finally 7-8. ACS patients are usually in hospital for 3 or 4 days provided there are no complications. It is therefore anticipated that days 0, 1-2 and 3-4 venesections may be performed whilst patient-participants are within the cardiology department. However an outpatient cardiology research clinic follow up will be arranged for day 7-8 to allow the final venesection for EPC analysis.

This pilot study will assess EPC response in patients that are able to undergo coronary intervention as part of their normal clinical management under current guidelines regardless of pre-existing comorbidities. The research team believe this will allow representation of "real world" patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with an acute coronary syndrome
* Are statin naive or receiving a statin other than atorvastatin, or atorvastatin at a dose less than 80mg daily
* Are able to give informed consent
* Have undergone coronary angiography/plasty
* Are able to attend follow up visits

Exclusion Criteria:

* Atorvastatin is contraindicated (e.g. allergic to excipient)
* Women of child bearing potential unless they are using a recognised effective form of contraception or are not sexually active and have no intention of becoming sexually active during the course of the trial
* Women who are breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Number of EPCs (per microliter of blood) in patient-participants admitted with an ACS loaded with atorvastatin 80 mg | 8 days
Number of EPCs (per microliter of blood) in patient-participants with different comorbid conditions | 8 days
Number of EPCs (per microliter of blood) in participants who have been loaded or reloaded with atorvastatin | 8 days
The time of onset of pain to loading/reloading strategies. | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Butler, Principal Investigator — University Hospitals of North Midlands NHS Trust
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No